CLINICAL TRIAL: NCT04747236
Title: A Randomized, Phase IIB, Multicenter, Trial of Oral Azacytidine Plus Romidepsin Versus Investigator's Choice in Patients With Relapse or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: Randomized Phase IIB Trial of Oral Azacytidine Plus Romidepsin Versus Investigator's Choice in PTCL
Acronym: PTCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Craig A Portell, MD, Professor of Medicine, Section Head for Hem Malignancies, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-001; FD-R-006814-01 (Other Grant/Funding Number: Office of Orphan Products Development (OOPD))
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PTCL
MeSH Terms: interventions — Azacitidine; romidepsin; belinostat; 10-propargyl-10-deazaaminopterin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZA and ROMI (Experimental): Oral Azacytidine (AZA) (300 mg daily on days 1-14) plus Romidepsin (ROMI) (14 mg/m2 as an intravenous infusion over 4 hours +/- 30 minutes on days 8, 15 and 22 of a 35-day cycle.
  Interventions: Drug: Azacytidine; Drug: Romidepsin
- Investigator's Choice (Active Comparator): Investigator's choice to include: ROMI, 14 mg/m2 IV infusion on days 1, 8, and 15 of a 28 day cycle, belinostat,1000 mg/m2 IV infusion on days 1-5 every 21 days, pralatrexate, 30 mg/m2 IV push once weekly for 6 weeks of a 7-week treatment cycle, or gemcitabine, 1000 mg/m2 IV infusion on days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Romidepsin; Drug: Belinostat; Drug: Pralatrexate; Drug: Gemcitabine

INTERVENTIONS:
Drug: Azacytidine — Azacytidine, 300 mg po daily on Days 1-14
  Other Names: Vidaza
  Arms: AZA and ROMI
Drug: Romidepsin — Romidepsin, 14 mg/m2 as an intravenous infusion over 4 hours on Days 8, 15, and 22 of a 35-day cycle
  Other Names: Istodax
Drug: Belinostat — Belinostat, 1000 mg/m2 as an intravenous infusion over 30 minutes on Days 1-5 every 21 days.
  Other Names: Beleodaq
  Arms: Investigator's Choice
Drug: Pralatrexate — Pralatrexate, 30 mg/m2 as an intravenous infusion over a 3-5 minute push once weekly for 6 weeks of a 7 week treatment cycle.
  Other Names: Folotyn
  Arms: Investigator's Choice
Drug: Gemcitabine — Gemcitabine, 1000 mg/m2 as an intravenous infusion over 30 minutes on Days 1, 8, and 15 of a 28 day cycle.
  Other Names: Gemzar
  Arms: Investigator's Choice

SUMMARY:
The purpose of this study is to find out whether the combination treatment of romidepsin and oral azacytidine is safe and effective in patients with Peripheral T-Cell Lymphoma (PTCL). This study will compare the experimental combination treatment of romidepsin and oral azacytidine to single agent drugs already determined effective in patients with PTCL. For the purposes of this study, the single agent drugs already used to treat lymphoma are called investigator's choice (IC), meaning the investigator will choose which one of these drugs to administer. The IC drug options include romidepsin, belinostat, pralatrexate or gemcitabine given alone. Funding Source: FDA OOPD.

DETAILED DESCRIPTION:
Peripheral T-Cell Lymphoma (PTCL) is a rare and heterogeneous group of non-Hodgkin lymphoma (NHL) originating from mature (or post-thymic or 'peripheral') T- lymphocytes and NK cells. They are considered very aggressive and are often resistant to conventional chemotherapy.

This study employs a stratified randomization with equal allocation within strata of patients to receive oral 5-azacytidine (AZA) plus romidepsin (ROMI) versus pre-specified investigator choice (ROMI, belinostat, pralatrexate or gemcitabine), for the treatment of relapsed or refractory (R/R) PTCL. The dose and schedule of AZA/ROMI has been determined from a phase I clinical trial of the combination. The primary objective of this study is to estimate the progression free survival (PFS) among patients receiving the combination compared to single agent of choice.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Patients must have histologically confirmed relapsed or refractory peripheral T-cell lymphoma as defined by 2016 WHO criteria (Section 13.7), who have progressed following one line of prior systemic therapy.

1. Patients are required to have no more than 3 lines of prior therapy (with cytoreductive therapy [ex ICE, DHAP, etc.] followed by autologous stem cell transplant counting as one line of therapy). Patients are eligible if they have relapsed after prior autologous or allogeneic stem cell transplant.
2. Patients with anaplastic large cell lymphoma are required to have received brentuximab vedotin (Bv) prior to study enrollment.
3. Measurable Disease as defined in Section 8.1.3.1.
4. Age ≥18 years.
5. ECOG performance status ≤2
6. Patients must have adequate organ and marrow function as defined below:

   Absolute neutrophil count (ANC): ≥1000/mm3 (≥1000/dL); Platelets: > 75,000/mm3; Serum Creatinine:< 2 x ULN OR creatinine clearance >50 mL/min/for patients with creatinine levels above ULN; Bilirubin: ≤ 1.5 x ULN (except in patients with Gilbert's disease, where bilirubin to 4x ULN is allowed); AST and ALT: ≤ 2 x ULN OR ≤ 3 X ULN in presence of demonstrable liver involvement; Serum potassium: ≥ 3.8 mmol/L; Serum magnesium≥1.8 mg/dL.
7. Negative urine or serum pregnancy test for females of childbearing potential
8. All females of childbearing potential and male subjects must agree to use an effective method of contraception (see section 5.4 for more details)
9. Be willing and able to provide written consent or assent for the trial.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Diagnosis of patch/plaque stage mycosis fungoides
2. Prior Therapy: Prior exposure to any hypomethylating agent or any histone deacetylase inhibitor (ex: romidepsin, chidamide, belinostat, or vorinostat); exposure to chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
3. Systemic steroids that have not been stabilized to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs.
4. No other concurrent investigational agents are allowed within 2 weeks of enrollment.
5. Known central nervous system metastases, including lymphomatous meningitis
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Nursing women
8. Other active concurrent malignancy (except non-melanoma skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of the breast (DCIS or LCIS). If there is a history of prior malignancy, the patient must be disease-free for ≥ 3-years. Patients whose lymphoma has transformed from a less aggressive histology remain eligible.
9. Patients known to be Human Immunodeficiency Virus (HIV)-positive.
10. Patients with active Hepatitis A, hepatitis B, or hepatitis C infection.
11. Concomitant use of CYP3A4 inhibitors (see Section 13.3)
12. History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
13. Abnormal coagulation parameters (PT >15 seconds, PTT>40 seconds, and/or INR >1.5) unless related to ongoing anticoagulation treatment required by the patient.
14. Known or suspected hypersensitivity to azacitidine (or any excipients in the formulation) or mannitol.
15. Any known cardiac abnormalities such as:

    * Congenital long QT syndrome
    * QTc interval ≥ 500 millisecond (using the Fridericia formula)
    * Patients taking drugs leading to significant QT prolongation (See Section 13.2)
    * Myocardial infarction within 6 months of C1D1. [Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event, may participate];
    * Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min);
    * Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV (see Section 13.4) In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
    * An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
    * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Section 13.5) and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI;
    * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest;
    * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes;
    * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria; or
    * Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2028-06-02 (Estimated); Study Completion 2030-06-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Day of randomization to day of progression or death, whichever comes first; or date of last disease assessment or date of transition to other treatment for those without an event, up to 72 weeks.
  Difference in progression free survival in subjects treated with AZA/ROMI versus pre-specified investigator choice.

SECONDARY OUTCOMES:
Overall survival | Day of randomization to day of death, whichever comes first; or date of last contact for those without an event, up to 72 weeks.
  Difference in overall survival in subjects treated with AZA/ROMI versus pre-specified investigator choice.
Complete response rate | Day of first objective response to 8 weeks following last dose of study treatment
  Difference in complete response (CR) rate in subjects treated with AZA/ROMI versus pre-specified investigator choice, based on the Revised Criteria for Response Assessment.
Overall response rate | Day of first objective response to 8 weeks following last dose of study treatment
  Difference in overall response (OR) rate in subjects treated with AZA/ROMI versus pre-specified investigator choice, based on the Revised Criteria for Response Assessment.
Duration of response rate | Day of first objective response to day of progression or death, whichever comes first; or date of last disease assessment or date of transition to other treatment for those without an event, up to 72 weeks.
  Difference in duration of response (DOR) rate in subjects treated with AZA/ROMI versus pre-specified investigator choice, based on the Revised Criteria for Response Assessment.
Time to progression | Day of randomization to day of progression, or date of last disease assessment or date of transition to other treatment for those without an event, up to 72 weeks.
  Difference in time to progression in subjects treated wtih AZA/ROMI versus pre-specified investigator choice.
Frequency of adverse events | From time of informed consent until 90 days after the last day of study treatment for all adverse events or anytime for serious adverse events considered related to the study intervention, through study completion, an average of 18 months.
  Frequency of adverse events in subjects treated wtih AZA/ROMI versus prespecified investigator choice assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Portell, MD, Principal Investigator — University of Virginia
Locations (6):
- United States (6):
  - VA Long Beach Health Care System, Long Beach, California
  - Yale Cancer Center, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107